CLINICAL TRIAL: NCT03215316
Title: Screening Expiratory Flow Limitation by Flow-time Curve
Acronym: FLOWLY
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-098
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Expiratory flow limitation (EFL) is defined as a dynamic condition that expiratory flow cannot be further increased with higher expiratory driving pressure. Under mechanical ventilation, it can cause intrinsic positive end-expiratory pressure (PEEP) and dynamic hyperinflation, and be associated with worse clinical outcome. The detection of EFL however needs special maneuvers and offline analysis of flow-volume curves, which are infeasible in routine practice and cannot be used during real-time monitoring. The investigators propose a new and simple approach using flow derived parameters to detect EFL in real time without needing any intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, intubated or tracheostomized
2. Receiving invasive mechanical ventilation in assist/control mode with PEEP ≥ 5 cmH2O
3. Receiving continuous intravenous sedation
4. Displaying a monotonous regular breathing pattern with no obvious asynchrony

Exclusion Criteria:

1. Severe hypoxemia in baseline clinical ventilator settings (SpO2 < 90%)
2. Hemodynamic instability (mABP <60 mmHg, systolic arterial pressure >180 mmHg, heart rate <40/min or >150/min)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients in the intensive care unit (ICU) receiving mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Outcome (Presence / absence of EFL) will be determined by off-line analysis of recorded flow-volume loops during PEEP reduction. | 2 years

SECONDARY OUTCOMES:
Percentage of intrinsic PEEP caused by the EFL. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided